CLINICAL TRIAL: NCT04004845
Title: Effect of a Labor Induction Protocol on Vaginal Delivery Rate
Brief Title: Labor Protocol Study
Status: Terminated | Type: Observational
Why Stopped: Study was temporarily paused due to COVID19 and ultimately terminated at the discretion of the PI
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Peter S. Bernstein, Principal Investigator, Montefiore Medical Center
Other Study IDs: 2018-9662
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Vaginal Delivery; Labor; Induced; Birth
MeSH Terms: interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pregnant women: We are including only women who are age 18 or over, who have a single baby (not twins), with the baby's head down, and are between 36 weeks 6 days and 42 weeks 0 days of pregnancy.
  Interventions: Drug: Cytotec; Drug: oxytocin; Device: Cervical Foley Balloon

INTERVENTIONS:
Drug: Cytotec — Misoprostol 25mcg vaginal
  Other Names: misoprostol
Drug: oxytocin — Oxytocin 10 IU/ml Solution for infusion
  Other Names: Pitocin
Device: Cervical Foley Balloon — Cervical Foley will be inflated to 80cc

SUMMARY:
The goal of this study is to see if there is a better way to induce labor.

DETAILED DESCRIPTION:
This is quasi-experimental prospective cohort study with historical control to examine the efficacy of a new labor induction bundle. The prospective cohort will consist of all eligible nulliparous and multiparous patients admitted for induction; the historical control group will consist of all eligible nulliparous and multiparous patients admitted for induction between August 2019 and February 2020. Patients who are part of the prospective cohort who do not consent to the labor bundle due to personal or physician preferences will be included in secondary analyses as a contemporary control group, however the sample size of this group will not be determined in advance.

Objective: To assess if implementation of an evidence-based labor induction bundle will increase the rate of vaginal delivery within 24 hours.

Hypothesis: Implementation of a labor induction bundle would result in a 30% increase in the rate of vaginal delivery within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. Cephalic presentation
3. Gestational age 36 weeks 6 days- 42 weeks 0 days at initiation of induction of labor
4. Age 18 and over

Exclusion Criteria:

1. Preterm (less than 36 weeks 6 days) at initiation of induction of labor
2. Non-cephalic presentation
3. Major fetal anomalies or intrauterine fetal death
4. Bishop score more than 6 at initiation of induction of labor
5. Any contraindication to any agents in the induction protocol (i.e. prior cesarean delivery or myomectomy, three or more contractions per ten minute period averaged over 30 minutes at the initiation of induction of labor, low lying placenta).
6. Any contraindication to vaginal delivery
7. Latex allergic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women with a single baby who are having their labor induced.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Vaginal Deliveries | Within 24 hours
  Percent vaginal delivery within 24 hours of initiation of labor induction

SECONDARY OUTCOMES:
Percent of vaginal delivery within 12 hours of initiating induction | Within 12 hours
Percent of deliveries (vaginal or cesarean) within 12 hours of initiating induction | Within 12 hours
Percent of deliveries (vaginal or cesarean) within 24 hours of initiating induction | Within 24 hours
Rate of vaginal delivery | Within 4 days
Rate of cesarean delivery | Within 4 days
Rate of operative vaginal delivery | Within 4 days
For patients undergoing cesarean delivery, rate of each indication for cesarean delivery | Within 4 days
Incidence of chorioamnionitis | Within 4 days
Number of vaginal exams | Within 4 days
  mean, median
Incidence of spontaneous internal version to non-cephalic presentation | Within 4 days
Incidence of umbilical cord prolapse | Within 4 days
Incidence of postpartum hemorrhage | Within 7 days
Incidence of transfusion of blood products | Within 7 days
Incidence of Neonatal 5-minute APGAR score <7 | Within 4 days
Incidence of Umbilical cord pH < 7, <7.1, <7.2 | Within 4 days
Incidence of Neonatal NICU admission | Within 7 days
Patient satisfaction with induction and delivery process measured on a scale of 1-10 - immediate | During delivery hospitalization
  Will analyze mean, median. Scale 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. Minimum score 1, Maximum score 10. A score of 1 is considered a worse outcome (completely dissatisfied) and 10 is considered a better outcome (completely satisfied). A score of 5 is neutral.
Incidence of shoulder dystocia | Within 4 days
Incidence of birth injuries (eg. brachial plexus injuries, musculoskeletal injuries, etc). | Within 7 days
Number of attending physicians managing induction of labor | Within 4 days
Number of attending-to-attending hand-off's | Within 4 days
Number of resident-to-resident team hand-off's | Within 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bernstein, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Weiler Division / Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] How HY, Leaseburge L, Khoury JC, Siddiqi TA, Spinnato JA, Sibai BM. A comparison of various routes and dosages of misoprostol for cervical ripening and the induction of labor. Am J Obstet Gynecol. 2001 Oct;185(4):911-5. doi: 10.1067/mob.2001.117358. PMID 11641677
- [Background] Pimentel VM, Arabkhazaeli M, Moon JY, Wang A, Kapedani A, Bernstein PS, Tropper PJ. Induction of labor using one dose vs multiple doses of misoprostol: a randomized controlled trial. Am J Obstet Gynecol. 2018 Jun;218(6):614.e1-614.e8. doi: 10.1016/j.ajog.2018.03.034. Epub 2018 Mar 31. PMID 29614276
- [Background] Macones GA, Cahill A, Stamilio DM, Odibo AO. The efficacy of early amniotomy in nulliparous labor induction: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):403.e1-5. doi: 10.1016/j.ajog.2012.08.032. Epub 2012 Aug 24. PMID 22959833
- [Background] Wei S, Wo BL, Qi HP, Xu H, Luo ZC, Roy C, Fraser WD. Early amniotomy and early oxytocin for prevention of, or therapy for, delay in first stage spontaneous labour compared with routine care. Cochrane Database Syst Rev. 2013 Aug 7;2013(8):CD006794. doi: 10.1002/14651858.CD006794.pub4. PMID 23926074
- [Background] Battarbee, A.N., Maternal and neonatal outcomes associated with early amniotomy in term nulliparous labor induction. Am J Obstet Gynecol, 2019. 220: p. 1.
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] Mackeen AD, Durie DE, Lin M, Huls CK, Qureshey E, Paglia MJ, Sun H, Sciscione A. Foley Plus Oxytocin Compared With Oxytocin for Induction After Membrane Rupture: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):4-11. doi: 10.1097/AOG.0000000000002374. PMID 29215519
- [Background] Schoen CN, Saccone G, Backley S, Sandberg EM, Gu N, Delaney S, Berghella V. Increased single-balloon Foley catheter volume for induction of labor and time to delivery: a systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2018 Sep;97(9):1051-1060. doi: 10.1111/aogs.13353. Epub 2018 Apr 25. PMID 29607491
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. Association of Early Amniotomy After Foley Balloon Catheter Ripening and Duration of Nulliparous Labor Induction. Obstet Gynecol. 2016 Sep;128(3):592-597. doi: 10.1097/AOG.0000000000001563. PMID 27500341
- [Background] Yee LM, Sandoval G, Bailit J, Reddy UM, Wapner RJ, Varner MW, Caritis SN, Prasad M, Tita ATN, Saade G, Sorokin Y, Rouse DJ, Blackwell SC, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Maternal and Neonatal Outcomes With Early Compared With Delayed Pushing Among Nulliparous Women. Obstet Gynecol. 2016 Nov;128(5):1039-1047. doi: 10.1097/AOG.0000000000001683. PMID 27741203
- [Background] Cahill AG, Srinivas SK, Tita ATN, Caughey AB, Richter HE, Gregory WT, Liu J, Woolfolk C, Weinstein DL, Mathur AM, Macones GA, Tuuli MG. Effect of Immediate vs Delayed Pushing on Rates of Spontaneous Vaginal Delivery Among Nulliparous Women Receiving Neuraxial Analgesia: A Randomized Clinical Trial. JAMA. 2018 Oct 9;320(14):1444-1454. doi: 10.1001/jama.2018.13986. PMID 30304425
- [Background] Simpson LL, Rochelson B, Ananth CV, Bernstein PS, D'Alton M, Chazotte C, Lavery JA, Zielinski K; Safe Motherhood Initiative Severe Hypertension in Pregnancy Work Group. Safe Motherhood Initiative: Early Impact of Severe Hypertension in Pregnancy Bundle Implementation. AJP Rep. 2018 Oct;8(4):e212-e218. doi: 10.1055/s-0038-1673632. Epub 2018 Oct 11. PMID 30319925
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430